CLINICAL TRIAL: NCT01172652
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Ziprasidone in Bipolar Disorder With Comorbid Lifetime Panic or Generalized Anxiety Disorder
Brief Title: Ziprasidone in Bipolar Disorder With Comorbid Lifetime Panic or Generalized Anxiety Disorder(GAD)
Acronym: PfizerAnxty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Pfizer (Industry); University of South Florida (Other); Lindner Center of HOPE (Other)
Responsible Party: Principal Investigator, patricia suppes, Director, Bipolar and Depression Research Program, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUP0005-17504
Record Dates: First submitted 2010-04-16; First posted 2010-07-30 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: Bipolar disorder; Anxiety; Panic; GAD; Generalized Anxiety Disorder
MeSH Terms: conditions — Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder; Anxiety Disorders | interventions — ziprasidone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ziprasidone (Experimental): Ziprasidone in the form of 40 and/or 80 mg capsules. Dose range: 40 to 160 mg/day.
  Interventions: Drug: Ziprasidone
- Placebo (Placebo Comparator): Administered in capsules identical to the ziprasidone capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — The minimum dose during study participation will be 40 mg/day, and the maximum dose allowed will be 160 mg/day.
  Other Names: Geodon; Zeldox
  Arms: ziprasidone
Drug: Placebo — Inactive control
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of ziprasidone monotherapy in comparison to placebo in the treatment of ambulatory bipolar disorder with co-morbid lifetime panic disorder or generalized anxiety disorder and current at least moderately severe anxiety.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel-group, 8-week trial of ziprasidone compared to placebo in outpatient subjects with a lifetime bipolar I, II, or NOS disorder, a lifetime panic or generalized anxiety disorder, and current diagnosis at least moderately severe anxiety symptoms. Approximately 50 subjects will be randomized. Subjects will be randomized to ziprasidone or placebo in a 1:1 ratio. No concomitant psychotropic medication will be allowed throughout the study except for prn lorazepam during the first two weeks for the management of affective and anxiety symptoms, prn zolpidem and zaleplon for the management of insomnia and benztropine for the management of EPS. Throughout the study, psychiatric scales will be used to assess psychiatric symptoms and the presence of treatment-emergent adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 and not older than 65.
* Subjects must have lifetime bipolar I, II, or NOS disorder as defined by DSM-IV TR criteria (26).
* Subjects must have lifetime panic disorder or generalized anxiety disorder (GAD) as defined by DSM-IV criteria (except clause "does not occur exclusively during a mood disorder" of Criterion F for GAD).
* Subjects' bipolar symptoms must be no more than moderate in severity, defined as a CGI-BP< 4 (27).
* Subjects' anxiety symptoms must be at least moderate in severity, defined as a CGI-S > 4 (28).
* Subjects must not be receiving regular mood stabilizing, antidepressant, antipsychotic, or anxiolytic medication for at least one week prior to baseline. Patients receiving fluoxetine or depot antipsychotics should be off these medications for at least four weeks prior to baseline.
* Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained.
* If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, barrier methods, intrauterine device) for at least one month prior to study entry and throughout the study.

Exclusion Criteria:

* Subjects who do not have lifetime bipolar disorder by DSM-IV-TR criteria (26).
* Subjects who do not have lifetime panic disorder or GAD by DSM-IV-TR criteria (26).
* Subjects who are receiving treatment with an anti-manic or mood stabilizing medication (lithium, valproate, carbamazepine, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication.
* Subjects whose bipolar symptoms are presently more than moderately severe (CGI-BP > 5) (27).
* Subjects whose anxiety symptoms are presently less than moderately severe (CGI-S < 3) (28).
* Subjects with clinically significant suicidal or homicidal ideation.
* Subjects with a current DSM-IV TR Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV TR diagnosis of a substance dependence disorder within the past six months; a lifetime DSM-IV TR psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
* Subjects with serious general medical illnesses as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
* Subjects with a clinically significant abnormality in their pre-study physical exam, vital signs, EKG, or laboratory tests.
* Subjects who are allergic to or who have demonstrated hypersensitivity or intolerance to ziprasidone.
* Women who are pregnant or nursing.
* Subjects who have received an experimental drug or used an experimental device within 30 days.
* Subjects who have a history of neuroleptic malignant syndrome.
* A patient with diabetes mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrollment glycosylated hemoglobin (HbAlc) >8.5%
  * Admitted to hospital for treatment of DM or DM related illness within the past 12 weeks
  * Not under physician care for DM
  * Physician responsible for patient's DM care has not indicated that the DM is controlled
  * Physician responsible for patient's DM care has not approved the patient's participation in the study
  * Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks before randomization. For thiazolidinediones(glitazones)this period should not be less than 8 weeks before randomization.
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks

Note: If a patient with DM meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Suppes, MD, PhD, Principal Investigator — VA Palo Alto Health Care System & Stanford School of Medicine
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System & Stanford School of Medicine, Palo Alto, California
  - University of South Florida Institute for Research in Psychiatry, Tampa, Florida
  - Lindner Center of Hope University of Cincinnati Medical Center, Mason, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suppes T, McElroy SL, Sheehan DV, Hidalgo RB, Cosgrove VE, Gwizdowski IS, Feldman NS. A randomized, double-blind, placebo-controlled study of ziprasidone monotherapy in bipolar disorder with co-occurring lifetime panic or generalized anxiety disorder. J Clin Psychiatry. 2014 Jan;75(1):77-84. doi: 10.4088/JCP.12m08297. PMID 24345758
- See also: Bipolar and Depression Research Program — http://bipolarresearch.stanford.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ziprasidone | Placebo
Started | 25 | 24
Completed | 6 | 17
Not Completed | 19 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (17.7) | 34.6 (12.2) | 36.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Clinician Global Improvement Scale (CGI-21)
Description: CGI-21 Anxiety Scale ranges from -10 (Very Bad. Could not be worse) to +10 (Major Improvement. Back to normal self).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 7.8 (1.7) | 3.4 (4.5)

2. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: Scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 10.2 (6.6) | 13.1 (10.4)

3. Secondary Outcome: Young Mania Rating Scale
Description: Four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. There are well described anchor points for each grade of severity. The authors encourage the use of whole or half point ratings once experience with the scale is acquired. Typical YMRS baseline scores can vary a lot. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 4.2 (5.1) | 4.4 (4.8)

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts. Usual cutoff points are: 0 to 6 - normal /symptom absent; 7 to 19 - mild depression; 20 to 34 moderate depression; >34 - severe depression.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 17.3 (11.5) | 19.1 (10.1)

5. Secondary Outcome: CGI-BP
Description: A guide for rating severity of manic and depressive episodes and the degree of change from the immediately preceding phase and from the worst phase of illness. Provides a set of instructions to facilitate the reliability of these ratings of mania, depression, and overall bipolar illness during treatment of an acute episode or in longer-term illness prophylaxis. Comprises two companion one-item measures evaluating the following:(a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale. The minimum value in each category is a score of 1 (indicating 'normal' or 'not ill') and the maximum value is a score of 7 (indicating 'very severely ill'). Higher scores indicate a worse outcome due to greater severity of bipolar symptoms. 1 = Very much improved 5 = Minimally worse 2 = Much improved 6 = Much worse 3 = Minimally improved 7 = Very much worse 4 = No change 3. Efficacy Index Rate this item on the basis of drug effect only.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 3.0 (1.5) | 3.0 (1.2)

6. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: A composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by panic, anxiety, phobic, or depressive symptoms. Patient rates the extent to which his or her 1) work, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. In each sector of the overall scale, the minimum score is a 1 (indicating that symptoms have been 'not at all' disruptive to functioning) and the maximum score is a 10 (indicating that symptoms have been 'extremely' disruptive to functioning). Each area of functioning is rated on a scale of 0 to either 3 or 5 (maximum score = 29-extreme vegetative state, minimum score = 0-person without disability) with the highest scores representing the higher level of disability. Higher scores indicate a worse outcome stemming from greater disability/impairment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 5 (4) | 9.9 (10.0)

7. Secondary Outcome: Sheehan Irritability Scale (SIS)
Description: SIS consists of seven items that assess symptoms of irritability, frustration, edginess/impatience, moodiness, anger with self, anger with others and temper during the previous week. Each item is assessed on an 11-point numeric rating scale ranging from 0 (not at all) to 10 (extremely). The SIS total score is calculated by summing of the scores for each of the seven individual items and ranges from 0 to 70. A higher score indicates a higher rate of irritability symptoms and therefore, a worse outcome.
Time Frame: 8 Weeks
Population: Outpatients with lifetime bipolar I disorder, bipolar II disorder, or bipolar disorder NOS by DSM-IV-TR criteria (26), who have co-morbid lifetime panic or generalized anxiety disorder, whose bipolar symptoms are no worse than moderately severe, and whose anxiety symptoms are currently at least moderately severe.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 25 | 24
Participants | 25 | 24

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the whole duration of the study which was 4/10 until 6/16. Each participant's adverse events were collected during the period of their participation up to
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone (N=25) | Placebo (N=24)
Hospitilazation (Social circumstances) | 0 (0) | 1 (1) — Illness related violence
Increase mood symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety, depression, possible suicide risk

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No